CLINICAL TRIAL: NCT01597375
Title: Therapeutic Control of Aspirin-Exacerbated Respiratory Disease (Aspirin)
Acronym: Aspirin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elliot Israel, MD (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor-Investigator, Elliot Israel, MD, Director of the Asthma Research Center, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2010P002961
Record Dates: First submitted 2012-04-30; First posted 2012-05-14 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Asthma, Aspirin-Induced; Aspirin Exacerbated Asthma
Keywords: Aspirin; Prasugrel; Asthma; AERD; Aspirin challenge; Aspirin desensitization; Aspirin induced asthma
MeSH Terms: conditions — Asthma, Aspirin-Induced; Asthma | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo then Prasugrel (Experimental): Subjects with AERD first received placebo oral tablet for 4 weeks prior to their aspirin challenge/desensitization. After aspirin challenge/desensitization subjects were discharged to home to washout the study drug from the first treatment phase. At the end of the 2-week washout period, subjects crossed over to the alternate treatment for 4 weeks of Prasugrel oral tablets [ (5 mg (for patients <60kg) or 10mg (> 60kg) daily, following a 60mg loading dose)] and returned for the second aspirin challenge.
  Because no period effect was observed, data obtained from all subjects while on placebo from either visit 2 or 3 were combined.
  Interventions: Drug: Placebo Oral Tablet; Drug: Prasugrel Oral Tablet
- Prasugrel then Placebo (Experimental): Subjects with AERD first received prasugrel oral tablets [ (5 mg (for patients <60kg) or 10mg (> 60kg) daily, following a 60mg loading dose)] prior to their aspirin challenge/desensitization. After aspirin challenge/desensitization subjects were discharged to home to washout the study drug from the first treatment phase. At the end of the 2-week washout period, subjects crossed over to the alternate treatment for 4 weeks of Placebo oral tablet.
  Because no period effect was observed, data obtained from all subjects while on Prasugrel from either visit 2 or 3 were combined.
  Interventions: Drug: Placebo Oral Tablet; Drug: Prasugrel Oral Tablet

INTERVENTIONS:
Drug: Placebo Oral Tablet — Participants will take a 60 mg loading dose. After they will take 10 mg by mouth daily if they weigh >60kg or 5 mg by mouth daily if they weigh <60 kg. They will take the drug for 4 weeks prior to the aspirin challenge/desensitization.
  Other Names: Placebo
Drug: Prasugrel Oral Tablet — Participants will take a 60 mg loading dose. After they will take 10 mg by mouth daily if they weigh >60kg or 5 mg by mouth daily if they weigh <60 kg. They will take the drug for 4 weeks prior to the aspirin challenge/desensitization.
  Other Names: Effient

SUMMARY:
The investigators are doing this research study to find out if giving a drug called prasugrel, which is used to prevent blood clots, can reduce reactions to aspirin in people with aspirin exacerbated respiratory disease (AERD), and to learn why taking aspirin every day can work as a treatment for people with AERD. People with AERD have symptoms of asthma, severe runny nose, polyps in the nose, and develop allergic reactions if they take medications like aspirin.

People with AERD can be desensitized to aspirin in order to be able to safely use it daily, but the investigators do not know if prasugrel may prevent reactions to aspirin and provide a safer way for people with AERD to tolerate aspirin.

The investigators also want to understand what is different about the cells and urine from subjects who have AERD, in comparison to subjects who have asthma but do not have AERD and subjects who have allergic rhinitis but do not have asthma. Lastly, the investigators want to understand how aspirin acts differently in subjects who have AERD, in comparison to subjects who have asthma but do not have AERD.

ELIGIBILITY:
Inclusion Criteria for Participants with AERD:

* History of physician-diagnosed asthma
* History of nasal polyposis
* History of at least one clinical reaction to oral aspirin or other nonselective COX inhibitor with features of both lower (cough, chest tightness, wheezing, dyspnea) and upper (rhinorrhea, sneezing, nasal obstruction, conjunctival itching and discharge) airway involvement.
* Stable asthma (post-bronchodilator FEV1 of 70% or better, no increase in baseline dose of oral glucocorticoids for at least 3 months, and no history of hospitalization or emergency room visits for asthma for at least the prior 6 months).
* No current smoking, defined as no daily tobacco smoking for at least 6 months and not more than one instance of tobacco smoking in the last 3 months.
* Non-pregnant
* Only those individuals who would otherwise meet clinical qualifications for aspirin desensitization and treatment with high-dose aspirin will be considered for enrollment in the study.

Inclusion Criteria for Participants who are Aspirin Tolerant Asthmatics:

* History of physician-diagnosed asthma.
* No current nasal polyposis confirmed by nasal examination.
* No history of any adverse reaction to aspirin or a COX inhibitor.
* Stable asthma (post-bronchodilator FEV1 of 70% or better, no increase in baseline dose of oral glucocorticoids for at least 3 months, and no history of hospitalization or emergency room visits for asthma for at least the prior 6 months).
* No current smoking
* Non-pregnant

Inclusion Criteria for Non Asthmatics with Allergic Rhinitis:

* No history of physician-diagnosed asthma.
* No current nasal polyposis confirmed by nasal examination.
* No history of any adverse reaction to aspirin or a COX inhibitor.
* No current smoking
* Non-pregnant
* Clinical history of symptoms consistent with allergic rhinitis and previously documented allergy to at least one environmental,immunoglobulin E (IgE) testing).
* Normal lung function (baseline FEV1 of 80% of predicted or better).
* A score of 4 or below on the Asthma Screening Questionnaire (33) and negative responses to asthma history questions

Exclusion Criteria for participants with AERD:

* Current breastfeeding
* History of bleeding diathesis or current use of anticoagulant or antiplatelet drugs
* Hypersensitivity to montelukast or thienopyridines
* History of peptic ulcer disease or gastrointestinal bleed
* Current severe gastro-esophageal reflux disease (GERD), defined as patient currently requiring more than 2 total doses of medication per day to treat persistent symptoms: either more than 2 doses of any single medication type (antacid, proton pump inhibitor, or H2 receptor antagonist), or more than 2 types of medication per day to treat symptoms
* History of systemic or life-threatening respiratory reaction to aspirin requiring intubation or administration of adrenalin
* Current use of any oral beta blocker (due to the risk of bronchospasm associated with beta blockers).
* History of transient ischemic attack or stroke, or diabetes.
* Current presence of uncontrolled hypertension.
* History of hepatic impairment or alcoholism, or evidence of abnormal liver function at Screening Visit. Aspartate transaminase (AST) and alanine transaminase (ALT) levels may not exceed 1.5x the upper limit of normal at Screening Visit (AST may not exceed 52 IU/L, ALT may not exceed 78 IU/L).

Exclusion Criteria for Participants with Aspirin Tolerant Asthma and Non Asthmatics with Allergic Rhinitis:

* Current breastfeeding
* History of bleeding diathesis or current use of anticoagulant or antiplatelet drugs
* Hypersensitivity to montelukast or thienopyridines
* History of peptic ulcer disease or gastrointestinal bleed
* Current severe GERD
* Current use of any oral beta blocker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-08-31 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital; Joshua Boyce, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Asthma Research Center, Boston, Massachusetts, United States

REFERENCES:
- See also: Click here for more info. — http://aerd.partners.org/research-studies/clinical-trial-therapeutic-control-of-aspirin-exacerbated-respiratory-disease/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 potential participants were screened at Brigham and Women's Hospital.
Pre-assignment Details: 46 of whom underwent randomization per protocol, and 40 of whom completed the trial and were analyzed.
Period: First Intervention (4 Weeks)
Arm/Group | Placebo Then Prasugrel | Prasugrel Then Placebo
Started | 23 | 23
Completed | 21 | 22
Not Completed | 2 | 1
Not completed — Uncontrolled Asthma | 1 | 0
Not completed — Needed surgery | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Washout (2 Weeks)
Arm/Group | Placebo Then Prasugrel | Prasugrel Then Placebo
Started | 21 | 22
Completed | 20 | 22
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Second Intervention
Arm/Group | Placebo Then Prasugrel | Prasugrel Then Placebo
Started | 20 | 22
Completed | 19 | 21
Not Completed | 1 | 1
Not completed — Failed to react at both Aspirin | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Prasugrel or Placebo oral tablets and who successfully completed both treatment assignments.
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Difference in PD2 (Provocative Dose of Aspirin That Elicits an Increase in Nasal Symptom Score of 2 During an Aspirin Challenge) on Prasugrel Versus Placebo
Description: The PD2 is the provocative dose of aspirin that elicits an increase in nasal symptom score of 2 during an aspirin challenge. The PD2 is calculated by:
  inverse〖log〗_10 (((2-(PrevTNSS-BaselineTNSS))×(〖log〗_10 ProvocDose-〖log〗_10 PrevDose))/((MaxTNSS-BaselineTNSS)-(PrevTNSS-BaselineTNSS) )+(〖log〗_10 PrevDose))
Time Frame: Difference in PD2 (provocative dose of aspirin that elicits an increase in nasal symptom score of 2 during an aspirin challenge) between Visits 2 and 3 (weeks 8 and 14), calculated at visit 3
Measure: Mean (Standard Error); unit: mg
Groups:
- Placebo: Subjects with AERD who received placebo oral tablets either the first or last 4 weeks of the study.
- Prasugrel: Subjects with AERD who received prasugrel oral tablets either the first or last 4 weeks of the study.
Arm/Group | Placebo | Prasugrel
Number analyzed (Participants) | 43 | 42
mg | 79 (15) | 139 (32)

2. Primary Outcome: Change From Baseline Expression Levels of COX-2 Transcript and Protein in Peripheral Blood Leukocytes of Subjects With AERD After 8 Weeks of Treatment With Aspirin.
Description: This study will compare this outcome within each participant between baseline (established at Visit 1, prior to initiation of prasugrel therapy) and at the completion of 8 weeks of aspirin therapy.
Time Frame: Evaluated at visits 1 and 4 (weeks 4 and 22)
Population: The planned experimental protocol for COX-2 analysis at the lab bench was unsuccessful, therefore no data was collected for this Outcome Measure
Arm/Group | Placebo | Prasugrel
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Difference in Participant's Provocative Dose of Aspirin When Pretreated With Prasugrel Versus Placebo
Description: We will monitor the dose of aspirin at which the participant shows symptoms (increased discomfort, 15% drop in FEV1) during the aspirin challenge/desensitization. We will compare the provocative aspirin dose obtained from the aspirin challenge occurring after pretreatment with prasugrel to the dose obtained after pretreatment with placebo.
Time Frame: Evaluated at visits 2 and 3 (weeks 8 and 14)
Measure: Mean (Standard Error); unit: mg
Arm/Group | Placebo | Prasugrel
Number analyzed (Participants) | 43 | 42
mg | 109 (15) | 164 (31)

4. Secondary Outcome: Change in Total Nasal Symptom Score(TNSS)From Baseline to Peak During Aspirin Challenge on Placebo Versus Prasugrel.
Description: The primary outcome in Part 1 will be the maximum Total Nasal Symptom Score (TNSS) attained for subjects with AERD during the clinical reaction to aspirin challenge. The primary analysis will compare this outcome within each participant after treatment with prasugrel versus placebo. Nasal symptoms including congestion, rhinorrhea, runny nose, itchy nose, sneezing, itchy eyes, teary eyes, itchy ears/throat, and eye redness were assessed on a 0- to 5-point scale (0, none-5, very severe) in response to the provocative dose of aspirin during aspirin challenge/desensitization and summed together to generate the TNSS score (range 0-40).
Time Frame: Data obtained at visits 2 and 3 (weeks 8 and 14) and change calculated at visit 3
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Prasugrel
Number analyzed (Participants) | 43 | 42
units on scale | 7 (0.8) | 6.5 (0.8)

5. Secondary Outcome: Change in Urinary LTE4 During Aspirin Challenge on Placebo Versus Prasugrel
Description: We will compare the participant's Leukotriene E4 (LTE4) obtained from the aspirin challenge done after pretreatment with prasugrel, the aspirin challenge done after pretreatment with placebo.
Time Frame: Change from visits 2 at visit 3 (weeks 8, 14), calculated and reported at visit 3
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | Prasugrel
Number analyzed (Participants) | 43 | 42
percentage change from baseline | 37 (70) | 19 (48)

6. Secondary Outcome: Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) Measurement After Aspirin Desensitization and High Dose Aspirin Treatment at 8 Weeks
Description: We will note difference in the fractional exhaled nitric oxide (FeNO) obtained before any treatment ( baseline ) and after one day Aspirin desensitization followed by 8 weeks Aspirin treatment ( 650 mg oral aspirin tablet twice daily )
Time Frame: Evaluated at baseline and reported at 8 weeks
Population: This was assessed across all participants with no planned comparisons between placebo and prasugrel.
Measure: Mean (Standard Deviation); unit: parts per billion
Groups:
- Subjects With AERD Completing 8 Weeks of Aspirin Treatment: Subjects with AERD who underwent Aspirin desensitization and 8 weeks of Aspirin treatment ( 650 mg of Aspirin twice daily )
Arm/Group | Subjects With AERD Completing 8 Weeks of Aspirin Treatment
Number analyzed (Participants) | 42
parts per billion | 15.8 (5.8)

7. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-7 (ACQ-7) Score After Aspirin Desensitization and High Dose Aspirin Treatment at 8 Weeks
Description: We will note difference in the Asthma Control Questionnaire-7 (ACQ-7) score [ The ACQ has 7 questions on a 7-point scale (minimum score of 0=no impairment, maximum score of 6= maximum impairment)] obtained before any treatment ( baseline ) and after one day Aspirin desensitization followed by 8 weeks Aspirin treatment ( 650 mg oral aspirin tablet twice daily )
Time Frame: Evaluated at baseline and reported at 8 weeks
Population: This was assessed across all participants with no planned comparisons between placebo and prasugrel.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects With AERD Completing 8 Weeks of Aspirin Treatment
Number analyzed (Participants) | 42
score on a scale | -0.11 (0.11)

8. Secondary Outcome: Change From Baseline in Prostaglandin Metabolites (PGD-M) Measurement After Aspirin Desensitization and High Dose Aspirin Treatment at 8 Weeks
Description: We will note difference in the Prostaglandin metabolites (PGD-M) measurement obtained before any treatment ( baseline ) and after one day Aspirin desensitization followed by 8 weeks Aspirin treatment ( 650 mg oral aspirin tablet twice daily )
Time Frame: Evaluated at baseline and reported at 8 weeks
Population: This was assessed across all participants with no planned comparisons between placebo and prasugrel.
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Subjects With AERD Completing 8 Weeks of Aspirin Treatment
Number analyzed (Participants) | 42
ng/mg creatinine | -1.4957 (6.9651)

9. Other Pre Specified Outcome: Baseline Differences in Platelet Chemistry in Subjects With AERD Compared to Controls
Description: To determine if there are baseline differences in the percentages of activated platelets, platelet-leukocyte aggregates, or the plasma levels of soluble platelet products in subjects with AERD, compared to aspirin tolerant asthmatics (ATA) and non-asthmatic controls.
Time Frame: Evaluated at visit 1 (week 4)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Effect of Prasugrel on Platelet Chemistry in Subjects With AERD During Aspirin Challenge.
Description: To determine if treatment with prasugrel changes the baseline percentages of activated platelets or platelet-leukocyte aggregates or changes the plasma levels of soluble platelet products during clinical reaction to aspirin
Time Frame: Evaluated at visit 2 and 3 (week 8 and 14)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of patient enrollment through study completion, an average of 20 weeks.
Arm/Group | Placebo | Prasugrel
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 13/43 | 13/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Prasugrel (N=42)
Bruising (Blood and lymphatic system disorders) | 3 (3) | 12 (12)
Upper Respiratory Tract Infection/Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (7)
Worsening of Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Muscle injury/Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (2)
Throat Infection (Infections and infestations) | 1 (1) | 1 (1)
Accidental ingestion of NSAID (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Systematic Reaction to Aspirin Challenge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Finger tingling/Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Light-Headedness (Nervous system disorders) | 1 (1) | 0 (0)
Lower leg edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mood Change (Psychiatric disorders) | 1 (1) | 0 (0)
Spider Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Viral Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No